CLINICAL TRIAL: NCT03539926
Title: Randomized, Controlled and Opened Trial on the Impact of the Use of a pH-Meter on the Domiciliary Control of the Urinary pH as Adjuvant to the Treatment of Cystinuric Patients
Brief Title: This Study Evaluates the Superiority of Daily Self-pH Monitorization of Lit-control®pH Meter Compared to the Monitorization of Reactive Strips (Standard of Care).
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Devicare S.L. (Industry)
Collaborators: Clever Instruments S.L. (Industry); Fundacio Puigvert (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: DEV-LCD-01-17
Record Dates: First submitted 2018-03-23; First posted 2018-05-30 (Actual); Last update posted 2018-11-21 (Actual); Status verified 2018-11

CONDITIONS: Cystinuria
Keywords: Cystinuria; pH Control
MeSH Terms: conditions — Cystinuria

STUDY DESIGN:
Intervention Model Description: Patients will receive the product for home pH monitoring, but they will keep following the doctor's recommendations indicated in the usual clinical practice.
  The proportion of patients will be 1: 1 between the study group (Lit-control®pH Meter) and the control group (test strips).
Masking Description: The process of randomization, either device use or use of strips, will be masked until the moment it is delivered to the patient. The random assignment to each product will be made through lists created by an ad hoc computer program.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lit-control®pH Meter (Experimental): The control of the urinary pH will be carried out twice a day: with the first urine in the morning and in the evening-night (approximately every 12h and at the same time). Measurements will be performed using the Lit-control®pH Meter device.
  Interventions: Device: Lit-control®pH Meter
- Reactive strips (Placebo Comparator): The control of the urinary pH will be carried out twice a day: with the first urine in the morning and in the evening-night (approximately every 12h and at the same time). Measurements will be performed using the reactive strips.
  Interventions: Diagnostic Test: Reactive strips

INTERVENTIONS:
Device: Lit-control®pH Meter — Alkalinization products will be used as standard clinical practice together with the pH monitoring through the Lit-control®pH Meter.
  Arms: Lit-control®pH Meter
Diagnostic Test: Reactive strips — Alkalinization products will be used as standard clinical practice together with the pH monitoring through the reactive strips.
  Arms: Reactive strips

SUMMARY:
This study evaluates the superiority of daily self-pH monitorization of Lit-control®pH meter compared to the monitorization of reactive strips (standard of care).

DETAILED DESCRIPTION:
Cystinuria is a disease of autosomal recessive inheritance. This disease belongs to the so-called orphan diseases although its prevalence may change depending on the country.

It is known that urinary pH is a risk factor for the formation of cystine crystals because their solubility is pH-dependent. In different studies it has been shown that the solubility of cystine in urine increases when alkalinizing urinary pH, thus reducing the likelihood of crystal formation. Therefore, the control of urinary pH along with hygienic-dietetic measures that alkalize the urine or decrease the urinary concentration of cystine (abundant intake of water, food, etc.) are highly recommended as a preventive method to prevent the formation of cystine crystals whose retention and growth results in the formation of stones.

The Lit-control®pH Meter is a pH meter that allows a patient to self-monitor its urinary pH in a comfortable and simple way. With this tool the patient is able to know if his urinary pH is within the recommended limits. In other medical fields it has been observed that home monitoring of clinically relevant physiological parameters is a way of empowering the patient that can positively affect their attitudes and behaviors (adherence to received treatment, quality of life) and potentially improve their medical condition. Specifically, in patients with chronic diseases, the self-monitoring has been associated with a significant reduction in hospitalizations and hospital readmissions.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old.
* Cystinuric patients, with or without urinary lithiasis at the time of inclusion.
* Patients who accept their participation in the study and give their informed consent.

Exclusion Criteria:

* Patients with pathologies that require pH control other than the one established in the study protocol to avoid the formation of kidney stones.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-04-09 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Percentage of days with pH levels within range 7 and 8, during 6 months of home self-monitoring. | 183 measurements (morning) in 6 months.
  Urinary pH measurement
Percentage of days with pH levels within range 7 and 8, during 6 months of home self-monitoring. | 183 measurements (afternoon) in 6 months.
  Urinary pH measurement
Measurement of the volume of crystalluria. | 1 measurement at the moment of enrollment
  volume of crystalluria
Measurement of the volume of crystalluria. | 1 measurement at 6 months
  volume of crystalluria
Blood: DNA extraction. | 1 measurement at the moment of enrollment
  Extraction of DNA for genetic study of mutations for cystinuria.
Sediment analysis for the determination of urinary infection. | 1 measurement at the moment of enrollment
  Sediment analysis for the determination of Ulcer Index (UI)
Sediment analysis for the determination of urinary infection. | 1 measurement at 6 months
  Sediment analysis for the determination of UI
Total time within the margins established as safe in the pH control (months). | 1 measurement through study completion [up to 6 months]
  Amount of time within the pH margins established as safe
Adherence level in pH measurements | Through study completion, fraction of pH measurements on the total possible. [up to 6 months]
  % compliance of the pH measurements
Adherence level to treatment | Through study completion, fraction of intakes on the total possible. [up to 6 months]
  % of the intakes of the medication.
Total number of adverse events reported. | Through study completion, number of events. [up to 6 months]
  Amount of adverse events reported
Blood Analysis. Glucose | Change from Baseline measurement at 6 months
  Glucose in mmol/L
Blood Analysis. Calcium phosphate | Change from Baseline measurement at 6 months
  calcium phosphate in µmol/L
Blood Analysis. Estimated Glomolecular Filtration Chronic Kidney Disease Epidemiology Collaboration (FG CKD-EPI) | Change from Baseline measurement at 6 months
  estimated FG CKD-EPI
Blood Analysis. Cystatin | Change from Baseline measurement at 6 months
  cystatin in mg/L (to be measured only if estimated FG> 45 or <ml /min / 1.73 m2 and albumin / creatinine in the urine <3 mg / mmol)
Blood Analysis. Creatinine | Change from Baseline measurement at 6 months
  creatinine in µmol/L
Blood Analysis. Urate | Change from Baseline measurement at 6 months
  urate in μmol/L
24h Urine Analysis. Weight | Change from Baseline measurement at 6 months
  Weight in kg
24h Urine Analysis. Size | Change from Baseline measurement at 6 months
  Size in m
24h Urine Analysis. Urinary volume | Change from Baseline measurement at 6 months
  Urinary volume in L
24h Urine Analysis. Calcium phosphate | Change from Baseline measurement at 6 months
  calcium phosphate in µmol/L
24h Urine Analysis. Citrate | Change from Baseline measurement at 6 months
  citrate in μmol/L
24h Urine Analysis. Urate | Change from Baseline measurement at 6 months
  urate in μmol/L
24h Urine Analysis. Magnesium | Change from Baseline measurement at 6 months
  magnesium in μmol/L
24h Urine Analysis. Sodium | Change from Baseline measurement at 6 months
  sodium in μmol/L
24h Urine Analysis. BMI | Change from Baseline measurement at 6 months
  weight and height will be combined to report BMI in kg/m^2
24h Urine Analysis. Potassium | Change from Baseline measurement at 6 months
  potassium in μmol/L
24h Urine Analysis. Urea | Change from Baseline measurement at 6 months
  urea in µmol/L
Urine for the study of crystalluria. Schedule | Change from Baseline measurement at 6 months
  First urine of the morning (totality) for the study of crystalluria. Patient will provide the last hour of urination and hour of urine obtention in the morning.
Urine for the study of crystalluria. Crystalline volume | Change from Baseline measurement at 6 months
  overall crystalline volume (μm3 / mL)
Urine for the study of crystalluria. Crystals | Change from Baseline measurement at 6 months
  type and number of crystals (crystals / μL)
Urine for the study of crystalluria. Urine volume | Change from Baseline measurement at 6 months
  urine volume in L
Urine for the study of crystalluria. pH | Change from Baseline measurement at 6 months
  pH
Urine for the study of crystalluria. Size | Change from Baseline measurement at 6 months
  size in μm
Urine for the study of crystalluria. Density | Change from Baseline measurement at 6 months
  Density in mg / mL.
Urine for the study of crystalluria. Aggregation | Change from Baseline measurement at 6 months
  aggregation
Urine for the study of crystalluria. Twinning | Change from Baseline measurement at 6 months
  twinning
Urine for the study of crystalluria. Quotient | Change from Baseline measurement at 6 months
  Quotient albumin / creatinine

SECONDARY OUTCOMES:
Sociodemographic and anthropometric questionnaire. | 1 day of enrollment
  Family and personal background and general data (sex, age, etc.).
Patient satisfaction questionnaire with the pH measurement method | 3 times in 6 months
  Visual Analogue Scale ranging from 1 (very dissatisfied) to 10 (very satisfied)
Physician satisfaction questionnaire with the pH measurement method | 3 times in 6 months
  Likert Scale with 4 categories: very dissatisfied, dissatisfied, satisfied, very satisfied

CONTACTS AND LOCATIONS:
Overall Officials: Oriol Angerri, MD, Principal Investigator — Fundacio Puigvert
Locations (1):
- Fundacio Puigvert, Barcelona, Spain